CLINICAL TRIAL: NCT00229736
Title: A Phase1 Open Label Safety Study of Intrastriatal Infusion of Adeno-Associated Virus Encoding Human Aromatic L-Amino Acid Decarboxylase (AAV-hAADC-2) in Subjects With Parkinson's Disease [AAV-hAADC-2-003]
Brief Title: A Study of AAV-hAADC-2 in Subjects With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAVhAADC2003
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AAV-hAADC-2 (9x10^10 vector genomes) (Experimental)
  Interventions: Genetic: AAV-hAADC-2
- AAV-hAADC-2 (3x10^11 vector genomes) (Experimental)
  Interventions: Genetic: AAV-hAADC-2

INTERVENTIONS:
Genetic: AAV-hAADC-2 — 9 x 10^10 vector genomes (vg) of AAV-hAADC-2 in a single dose of 200 µL bilaterally infused over 4 striatal targets
  Arms: AAV-hAADC-2 (9x10^10 vector genomes)
Genetic: AAV-hAADC-2 — 3 x 10^11 vector genomes (vg) of AAV-hAADC-2 in a single dose of 200 µL bilaterally infused over 4 striatal targets
  Arms: AAV-hAADC-2 (3x10^11 vector genomes)

SUMMARY:
Safety Study in subjects with Parkinson's Disease

DETAILED DESCRIPTION:
In a patient with Parkinson's disease, the part of the brain called the substantia nigra progressively loses the ability to send dopamine signals to the striatum.

To compensate for the loss of striatal dopamine, most patients take L-dopa, an approved drug which is converted to dopamine by an essential enzyme - AADC.

With time, however, the brain loses its remaining ability to convert L-dopa to dopamine and thus the drug becomes progressively less effective.

In the therapy being studied, the gene coding for the enzyme that converts L-dopa to dopamine (AADC) is inserted into a common, non-pathogenic virus (AAV) to which > 90% of humans have been exposed.

The AAV will help to transport the AADC into the brain cells.

AAV-hAADC-2, the investigational drug being studied, is injected into the striatum during a surgical procedure.

Patients who undergo the procedure would continue to take L-dopa; AAV-hAADC-2 is intended to provide, directly to the brain, the missing enzyme needed to convert L-dopa to dopamine.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent.
* Diagnosis of idiopathic Parkinson's disease (two of four cardinal features - tremor, bradykinesia, rigidity and postural instability - plus early dopaminergic responsiveness of symptoms and absence of any cardinal signs of more widespread neurological disease).
* Age ≤ 75 years.
* Age at diagnosis ≥ 40 years.
* Duration of levodopa therapy ≥ 5 years (number of years is cumulative since diagnosis, does not need to be continuous).
* Hoehn and Yahr Stage III to IV off medication at entry.
* Unified Parkinson's Disease Rating Scale (UPDRS), Part III, minimum motor score of 20 to a maximum motor score of 60 in the "OFF" state.
* Positive response to dopaminergic therapy as evidenced by a decrease in UPDRS motor scores between the defined "OFF" and "ON" states: a minimum of 8 points improvement in the UPDRS after dopaminergic therapy.
* Candidate for surgical therapy for Parkinson's disease because of intractable motor fluctuations, defined as a subscore on UPDRS Part IV section B ("Clinical Fluctuations" score of 3 (minimum) to 7 (maximum) during the "ON" state, not responsive to optimal medical therapy.
* MRI (magnetic resonance imaging)within the past two years and MRI does not show any conditions that are clinically significant with respect to risks for brain surgery.
* Subjects must agree to use barrier contraception, until three consecutive PCR (polymerase chain reaction) samples are negative, if the subject or partner is of childbearing potential.
* Must be able to comply with the requirements of the study, including the need for frequent and prolonged follow-up.
* Subjects must have been on both optimal and stable medications for treatment of their Parkinson's disease for at least two months prior to being eligible for participation in the study.
* Subjects must have baseline Hematology and Chemistry values within the normal laboratory ranges unless the out of range values are not clinically significant with respect to general surgery.

Exclusion Criteria:

* Unable or unwilling to meet requirements of the study.
* Atypical Parkinsonian syndromes due to drugs (e.g. metoclopramide, flunarizine), metabolic disorders (e.g. Wilson's disease), encephalitis, or degenerative diseases (e.g., juvenile Huntington's disease, progressive supranuclear palsy, multisystem atrophy, dementia with Lewy bodies).
* History of three (3) hours or more of intense or violent dyskinesias in the past six (6) months.
* Previous stereotactic neurosurgery for Parkinson's disease (pallidotomy, thalamotomy, deep brain stimulation).
* Mini-Mental™ State Examination (MMSE) < 26 or screening neuropsychological evaluation compatible with dementia.
* Hallucinations or delusions due to medication or underlying mental illness within 6 months of screening; documented history of schizophrenia or other psychotic disorder.
* History of serious mood disorder that, in the opinion of the Investigator, is not effectively managed.
* History of stroke or other currently significant or poorly controlled cardiovascular disease.
* Intracranial neoplasia, clinically significant neurological diseases (for example, significant brain atrophy not consistent with age).
* History of other malignancy, with the exception of treated cutaneous squamous cell or basal cell carcinoma, within 5 years.
* Uncontrolled hypertension: systolic blood pressure consistently >160 mmHg with no attempt at treatment.
* Coagulopathy or need for ongoing anticoagulant therapy.
* Clinically significant immune dysfunction (for example, those that require the use of immunosuppressive drugs).
* Geriatric Depression Scale (GDS; Mood Assessment Scale - Short Form) score of >10 or, if on anti-depressants, a score >5.
* Monoamineoxidase (MAO)inhibitors, and/or anti-psychotic medications.
* Contraindication to magnetic resonance imaging (MRI).
* Neutralizing antibody titer to AAV-2 ≥ 1:1200.
* For pre-menopausal women: a positive (+) urine pregnancy test.
* Dopaminergic blocking agents within 30 days prior to the Baseline visit.
* Investigational agents within 12 weeks prior to the Baseline visit.
* Clinically active infection with adenovirus or herpes virus.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of intrastriatal administration of AAV-hAADC-2 as measured by Adverse Events in subjects with mid- to late-stage Parkinson's Disease. | Time of treatment through Month 60.

SECONDARY OUTCOMES:
The effect of AAV-hAADC-2 on clinical status as recorded in subject diaries, by clinical assessment, and daily levodopa requirement. | Time of treatment through Month 60.
The relationship between the dose of AAV-hAADC-2 vector infused and the resulting level of striatal AADC expression by FMT-PET imaging. | Time of treatment through Month 60

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Christine CW, Starr PA, Larson PS, Eberling JL, Jagust WJ, Hawkins RA, VanBrocklin HF, Wright JF, Bankiewicz KS, Aminoff MJ. Safety and tolerability of putaminal AADC gene therapy for Parkinson disease. Neurology. 2009 Nov 17;73(20):1662-9. doi: 10.1212/WNL.0b013e3181c29356. Epub 2009 Oct 14. PMID 19828868